CLINICAL TRIAL: NCT05976230
Title: Special Drug Use Surveillance of Entresto Tablets (Hypertension, CLCZ696A1402): ENLIGHT
Brief Title: Special Drug Use Surveillance of Entresto Tablets (Hypertension)
Acronym: ENLIGHT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696A1402
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: hypertension; Entresto; Entresto Tablets; actual clinical practice; Japan; sacubitril/valsartan; sacubitril valsartan sodium hydrate
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Entresto: Patients administered Entresto by prescription
  Interventions: Drug: Entresto

INTERVENTIONS:
Drug: Entresto — There is no treatment allocation. Patients administered Entresto by prescription that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Entresto Tablets

SUMMARY:
This is a single arm, multicenter, observational study to evaluate the safety and efficacy of Entresto Tablets during the first 52 weeks of treatment in Japanese patients with hypertension.

DETAILED DESCRIPTION:
This study is a special drug use surveillance to collect information on the safety specifications under the actual clinical practice of Entresto Tablets in patients with hypertension in Japan to confirm the occurrence and timing of onset of events related to the safety specifications and investigate their risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given written consent to participate in this study before the start of treatment with Entresto
2. Patients who used Entresto for the first time for the indication of hypertension

Exclusion Criteria:

1. Patients who have received a formulation containing the same ingredient as Entresto (including investigational product or post-marketing clinical study drug)
2. The following patients for whom administration of Entresto is contraindicated in the package insert:

   * Patients with a history of hypersensitivity to any of the ingredients of Entresto
   * Patients who are receiving angiotensin-converting enzyme inhibitors (alacepril, imidapril hydrochloride, enalapril maleate, captopril, quinapril hydrochloride, cilazapril hydrate, temocapril hydrochloride, delapril hydrochloride, trandolapril, benazepril hydrochloride, perindopril erbumine, and lisinopril hydrate) or who discontinued these drugs within 36 hours.
   * Patients with a history of angioedema (angioedema due to angiotensin II receptor antagonists or angiotensin converting enzyme inhibitors, hereditary angioedema, acquired angioedema, idiopathic angioedema, etc.)
   * Patients with diabetes mellitus who are receiving aliskiren fumarate
   * Patients with severe hepatic impairment (Child-Pugh class C)
   * Pregnant or possibly pregnant women
3. Patients with a history or complication of cardiac failure
4. Patients who have been hospitalized at the start of treatment with Entresto

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese patients with hypertension using Entresto
Sampling Method: Non-Probability Sample
Enrollment: 1125 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with hypotension, hyperkalemia, and renal impairment/failure | Up to 52 weeks
  To investigate the safety of 52 weeks of treatment with Entresto in patients with hypertension in a real-world setting. In particular, the occurrence status of hypotension, hyperkalemia, and renal impairment/renal failure

SECONDARY OUTCOMES:
Percentage of patients with hypotension, hyperkalemia, and renal impairment/failure by risk factor | Up to 52 weeks
  To identify risk factors associated with the development of hypotension, hyperkalemia, and renal impairment/failure
Odds ratio (OR) for each risk factor of hypotension, hyperkalemia, and renal impairment/failure | Up to 52 weeks
  To identify risk factors associated with the development of hypotension, hyperkalemia, and renal impairment/failure
Change from baseline in sitting systolic blood pressure (sSBP) and sitting diastolic blood pressure (sDBP) over time | Up to 52 weeks
  To evaluate the efficacy of 52 weeks of treatment with Entresto in a real-world setting
Percentage of patients who achieved blood pressure control at each evaluation time point | Up to 52 weeks
  To evaluate the efficacy of 52 weeks of treatment with Entresto in a real-world setting
Percentage of patients who achieved improvement in sSBP and sDBP at each evaluation time point | Up to 52 weeks
  To evaluate the efficacy of 52 weeks of treatment with Entresto in a real-world setting

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (86):
- Japan (86):
  - Novartis Investigative Site, Anjo, Aichi-ken
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Kasugai, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Okazaki, Aichi-ken
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Yatomi, Aichi-ken
  - Novartis Investigative Site, Inzai, Chiba
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Sakura, Chiba
  - Novartis Investigative Site, Yotsukaidō, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Saijō, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Kasuya Gun, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Nakagawa, Fukuoka
  - Novartis Investigative Site, Omuta, Fukuoka
  - Novartis Investigative Site, Yame, Fukuoka
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Takehara, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kasai, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Bandō, Ibaraki
  - Novartis Investigative Site, Chikusei, Ibaraki
  - Novartis Investigative Site, Koga, Ibaraki
  - Novartis Investigative Site, Moriya, Ibaraki
  - Novartis Investigative Site, Ryūgasaki, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Aiko-gun, Kanagawa
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Yamaga, Kumamoto
  - Novartis Investigative Site, Iki, Nagasaki
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Nakatsu, Oita Prefecture
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Ikeda, Osaka
  - Novartis Investigative Site, Minoo, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Kashima, Saga-ken
  - Novartis Investigative Site, Kishima-gun, Saga-ken
  - Novartis Investigative Site, Tosu, Saga-ken
  - Novartis Investigative Site, Ureshino, Saga-ken
  - Novartis Investigative Site, Asaka, Saitama
  - Novartis Investigative Site, Fujimino, Saitama
  - Novartis Investigative Site, Gyōda, Saitama
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Niiza, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Satte, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Akishima, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Kokubunji, Tokyo
  - Novartis Investigative Site, Koto-ku, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
  - Novartis Investigative Site, Yamaguchi, Yamaguchi
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Saitama

IPD SHARING:
Plan to Share IPD: No